CLINICAL TRIAL: NCT06135857
Title: Electromuscular Stimulation Therapy as a Prophylactic Method to Reduce Thromboses Related to PICC Catheters in Patients Hospitalized in Critical Care Units. Randomized Clinical Trial.
Brief Title: Electromuscular Stimulation Therapy as a Prophylactic Method to Reduce Thromboses Related to PICC Catheters in Patients Hospitalized in Critical Care Units.
Acronym: ECOEMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta (Other)
Responsible Party: Principal Investigator, Gerez Acevedo, Principal Investigator, Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023.151
Record Dates: First submitted 2023-11-06; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Thrombosis; Catheter, Infusion Catheter (Vascular)
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Device: Protocol ECOEMS
- Control group (No Intervention)

INTERVENTIONS:
Device: Protocol ECOEMS — Use electo estimulation therapy. The 4-channel stimulator will be used. The 6 electrodes will be located on the biceps, triceps and deltoids. Two daily sessions will be distributed, five days a week, lasting 20 minutes, the vascular program designed by the electro stimulation team itself will be applied.
  Arms: Intervention group

SUMMARY:
Introduction: The placement of a peripheral inserted central catheter (PICC) is a common practice in the hospital setting. However, despite all the advances reported, venous devices are not free of complications and catheter-related thrombosis (CRT), being one of the most prevalent. Electro muscular stimulation therapy can be a measure for the prevention of CRT. Objective: To know the efficacy of electro muscular stimulation therapy in patients hospitalized in critical care units to prevent venous thrombosis related to PICC catheters. Methodology: A multicenter Randomized Clinical Trial (RCT) will be carried out at the Dr. Josep Trueta University Hospital in Girona, Hospital del Mar in Barcelona, Althaia Foundation in Manresa. With a total of 68 patients with PICC catheters in critical care units, they will be randomly assigned to the intervention group (n=34) to whom, in addition to the usual protocolized care related to the vascular catheter, will be applied e Eco-EMS protocol, or the control group (n=34) to which only the usual protocolized care related to the vascular catheter was applied. Intervention: It will consist of the application of electrostimulation therapy five days a week, two daily sessions of 20 minutes in the intervention group. Both groups underwent five ultrasound examinations after the placement of the PICC to determine the appearance of CRT. Expected results: It is expected to observe that the application of the Eco-EMS protocol reduces thrombosis in the patients of the intervention group, compared to those of the control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the critical unit with a PICC whose insertion is done by the EIAV of the same hospital.
* Patients between 18 and 80 years of age.
* Treatments related to the device protocolized by the same hospital as the EIAV implanter.

Exclusion Criteria:

* Patients who do not sign informed consent.
* Patients with pacemakers and/or implantable automatic defibrillators.
* Patients with epilepsy.
* Removal of the device within the first 15 days after insertion.
* Hospital discharge, transfer to another hospital or death lethalis during the duration of the study.
* Displacement of the tip of the catheter outside the lower ⅓ of the superior vein cava during the study period.
* Presence of lesions in the place where the electrodes must be placed to perform the electrostimulation therapy.
* Non-compliance with catheter monitoring: Of the five ultrasound controls protocolized in the study, 80% were not complied with.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
To know the effectiveness of electromuscular stimulation therapy in patients hospitalized in critical care units to prevent venous thrombosis related to PICC catheters. | 15 days
  Ultrasound will be used to measure whether or not there is the appearance of thrombosis related to the PICC catheter.

IPD SHARING:
Plan to Share IPD: Undecided